CLINICAL TRIAL: NCT00006232
Title: A Randomized Trial Comparing Z-Dex With VAD as Induction Therapy for Patients With Multiple Myeloma
Brief Title: Combination Chemotherapy in Treating Patients With Stage II or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West of Scotland Lymphoma Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: WSLG-H31; CDR0000068156 (Registry Identifier: PDQ (Physician Data Query)); EU-20032; ISRCTN65684689
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2007-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Doxorubicin; Idarubicin; Vincristine

INTERVENTIONS:
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: idarubicin
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective for multiple myeloma.

PURPOSE: This randomized phase III trial is comparing two combination chemotherapy regimens to see how well they work in treating patients with stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the partial and complete response rates in patients with multiple myeloma treated with induction therapy comprising idarubicin and dexamethasone vs vincristine, doxorubicin, and dexamethasone.
* Compare the disease progression, time to achieve maximal response, and duration of response in patients treated with these 2 regimens.
* Compare the quality of life of patients treated with these 2 regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral idarubicin and oral dexamethasone daily on days 1-4. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral dexamethasone daily on days 8-11 during course 1 only.
* Arm II: Patients receive oral dexamethasone daily, doxorubicin IV continuously, and vincristine IV continuously on days 1-4. Courses repeat as in arm I. Patients receive additional dexamethasone as in arm I.

Patients without a maximal response after completion of course 4 may receive up to 2 additional courses.

Quality of life is assessed at baseline and then prior to each study course.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 200 patients (100 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage II or III multiple myeloma

  * No prior therapy except local radiotherapy to bone lesions
* No indolent multiple myeloma
* No monoclonal gammopathy of unknown significance

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.34 mg/dL

Renal:

* No end stage renal failure (creatinine greater than 5.65 mg/dL after rehydration)
* No requirement for dialysis

Other:

* No other medical condition that would preclude intensive treatment
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Concurrent local radiotherapy allowed for painful lesions or lesions that appear likely to lead to an imminent fracture

Surgery

* See Disease Characteristics

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1996-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Comparison of response rates

SECONDARY OUTCOMES:
Time to achieve a maximal response
Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cook, MD, PhD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (12):
- United Kingdom (12):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Royal Liverpool and Broadgreen Hospitals NHS Trust, Liverpool, England
  - New Cross Hospital, Wolverhampton, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Vale Of Leven D G Hospital, Alexandria, Scotland
  - Dumfries Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland